## **Cover Page**

**Title**: Brief Protocol Summary-- Addressing Intersectional Stigma: Testing THRIVE 365 for Black Sexual Minority Men (On The Daily)

NCT Number: NCT05376397

**Document Date**: 12/18/2023

## **Brief Protocol Summary**

The sample consisted of Black sexual minority men (SMM) living with HIV and connected with the community-based organization, THRIVE SS. THRIVE SS is an Atlanta, GA based CBO that focuses on health equity for Black SMM, most of whom are living with HIV, through cultivating peer support, advocacy, and community building. The study team recruited a nonrandom purposive sample through advertisements on THRIVE SS's social media and email blasts. Eligibility criteria for this analysis were: 16 years old or older, identifying as masculine, identifying as Black/African American, reporting being attracted to and/or sexually active with men, able to complete all procedures in English, mobile access to the internet in order to complete the once-daily survey procedures. After the screening eligible for the study, participants received an invitation to participate in a HIPPA compliant WebEx informed consent meeting and baseline assessment with a trained research assistant. After baseline was a 14-day daily diary study with surveys administered on an Internet-based Qualtrics platform. Across all days, participants received 8 PM text-messages with links to their daily surveys. For those who had not completed the survey by 9:30 PM, they received an automatic reminder message. Surveys included measures of psychological and behavioral variables. We used simple randomization to vary the order of administration of all instruments. In line with a pre-post, one-arm trial, participants did not have access to the iTHRIVE 365 intervention for days 1-7 then received access to register and use the invention for days 8-14. The follow-up assessment occurred at the end of the 2week daily diary period. We collected summary paradata (i.e., process data detailing app usage) on intervention page access. Participants received \$30 for baseline and follow-up and \$1.50 per survey for the first 7 daily surveys and \$2.50 for the next 7 surveys, with a \$5 bonus for completing all surveys (total maximum: \$93). The Rutgers University institutional review board approved all study procedures.

iTHRIVE 365 is a multicomponent intervention that uses mHealth features in alignment with 4 community priorities identified in our formative CBPR research: (1) Support HIV and psychological health knowledge and motivation; (2) Foster a sense of community and positive social connections among Black SMM; (3) Connect users to Black SMM-affirming health care, including HIV treatment and mental health care; (4) Provide resources for housing, transportation, and other economic empowerment. In line with best-practices for administering and testing interventions with mHealth components with trials of intervention principles (TIPs), iTHRIVE 365 deploys intervention elements that contain content that may be updated to maintain user engagement, but ultimately serve to accomplish delineated intervention strategies that match the community priorities. iTHRIVE 365 uses these intervention elements: (1) Weekly HIV and psychological health information and motivation content and daily health notifications; (2) Online moderated forums, interpersonal chats, and community calendars; (3) Linkage to biopsychosocial health care via THRIVE SS's network of Black SMM-affirming providers; and (4) Housing and economic resources through THRIVE SS's direct support and referral network. The health knowledge and motivation content includes a health maintenance notification system and content covering HIV and psychological health content that are evidence-based and culturally-tailored by the

Rutgers School of Public Health and THRIVE SS team for Black SMM. The health maintenance notification system allows users to input the timing and dosage of medications or health practices (e.g., mindfulness meditation) to receive personalized reminders. Similar notification systems, such as automated pill reminders, have been shown to improve ART adherence. The HIV health content includes educational and motivational material developed by THRIVE SS that is supported by evidence-based HIV treatment approaches. The psychological health content includes psychoeducation and exercises from cognitive behavioral therapy (CBT), positive psychology (PPI), and dialectic behavioral therapies (DBT) aimed at promoting individual education and motivation and facilitating users to identify and replace negative thought and behavioral patterns consistent with a transtheoretical approach. In the pilot version of iTHRIVE 365 tested here, the health knowledge and motivation content was housed in the home/landing and pill reminder pages. The social support content includes a community calendar that provides up-to-date information on THRIVE SS-led and other Black SMM community events in the Atlanta, GA area and gives users the option to receive reminder notifications about them. It also includes evidence-based features such as a moderated forum with discussions on topics generated by THRIVE SS staff or proposed by users and approved by staff. These forums have supported discussions on topics such as confronting stigma, medication side effects, and shared interests in popular culture. In line with guidance from formative focus groups, the forums are meant to support community around more than just HIV (e.g., finances, music) and include community guidelines that require users to refrain from personal attacks, hateful language, and other forms of communication that may cause forums to be unsafe for users. Forum moderators are THRIVE SS staff who identify violations of community guidelines. The interpersonal chat is a private chat between users that is only restricted if a user reports a violation of community guidelines. In the pilot version of iTHRIVE 365 tested here, the social support content was housed in the community, calendar, and chat pages. The access to affirming health care feature allows users to request THRIVE SS institutional support including linkage to psychotherapy, Black SMM support groups, HIV care, and COVID care. THRIVE SS draws on a network of Black SMM-affirming Atlanta, GA-area health care providers that has been developed and vetted by THRIVE SS over 10 years through site visits and qualitative evaluations from staff and members that assess aspects of affirming contexts (e.g., ease of access, patient comfort, and provider cultural humility). Given the timing of the deployment of this version of iTHRIVE 365 first in 2021, we included a CDC COVID screener (https://www.cdc.gov/screening/index.html) in this section. The housing and economic empowerment resources linkage features allow users to request free transportation, food assistance, culturally-appropriate clothes, and connection to housing support.

empowerment resources linkage features allow users to request free transportation, food assistance, culturally-appropriate clothes, and connection to housing support. Transportation costs are covered through paid transit passes and direct cash assistance. Clothes and food assistance are provided on-site at THRIVE SS and through THRIVE SS partner organizations. Housing assistance is managed by THRIVE SS case workers and includes transitional housing at a THRIVE SS-owned transitional home that provides housing for up to 5 months for those seeking a permanent residence and referrals to housing vouchers and other housing support in THRIVE SS's network. In the pilot version of iTHRIVE 365 tested here, the access to affirming health care and economic empowerment features were housed in the linkage page.